CLINICAL TRIAL: NCT01165580
Title: Pharmacokinetics and Safety of Valganciclovir in Pediatric Heart Transplant Recipients < 4 Months of Age
Brief Title: A Study on the Pharmacokinetics and Safety of Valcyte (Valganciclovir) in Pediatric Heart Transplant Recipients Less Than 4 Months of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NP22523; 2010-021172-28
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cytomegalovirus Infections, Heart Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: valganciclovir [Valcyte]

INTERVENTIONS:
Drug: valganciclovir [Valcyte] — oral dose, Days 1 and 2

SUMMARY:
This open label study will assess the pharmacokinetics and the safety and tolerability of Valcyte (valganciclovir) powder for oral solution in neonatal and infant heart transplant patients < 4 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 0 to < 4 months (< 125 days) of age at the time of the last PK assessment in this study
* Parent or guardian of the patient is willing and able to give written informed consent
* Patient has received a first heart transplant
* Patient is at risk of developing cytomegalovirus (CMV) disease and is being treated with i.v. ganciclovir or oral valganciclovir for prevention of CMV
* Adequate hematological and renal function
* Able to tolerate oral medication (any appropriate form of tube feeding is acceptable)

Exclusion Criteria:

* Allergic or significant adverse reaction to acyclovir, valacyclovir or ganciclovir in the past
* Severe, uncontrolled, clinically abnormal diarrhea
* Liver enzyme elevation of more than five times the upper limit of normal for AST (SGOT) or ALT (SGPT)
* Patient requires use of any protocol prohibited concomitant medications
* Patient has previously participated in this clinical trial

Max Age: 124 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration versus time curve of ganciclovir | 0, 1-3, 3-7, 7-12, 24 hours post-dose
Apparent volume of distribution of ganciclovir | 0, 1-3, 3-7, 7-12, 24 hours post-dose
Terminal half-life of ganciclovir | 0, 1-3, 3-7, 7-12, 24 hours post-dose
Peak concentration of ganciclovir | 0, 1-3, 3-7, 7-12, 24 hours post-dose

SECONDARY OUTCOMES:
Safety (Incidence of adverse events) | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (16):
  - Loma Linda, California
  - Palo Alto, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - The Bronx, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Edmonton, Alberta, Canada
- Madrid, Madrid, Spain